CLINICAL TRIAL: NCT06905899
Title: Effect of Audio Book Applıcatıon on Patıents Blood Pressure, Pulse Rate and Anxıety Levels Before Total Knee Replacement Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beyza Yilmaz (Other)
Responsible Party: Sponsor-Investigator, Beyza Yilmaz, principal investigator, Ahi Evran University Education and Research Hospital
Organization: Ahi Evran University Education and Research Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: AhiEvranUERHseslikitap1487
Record Dates: First submitted 2025-02-19; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stress
Keywords: anxiety; blood pressure; before surgery; total knee prosthesis; audio book
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study will be conducted for 2 groups as experimental and control groups.
Masking Description: The researcher applied forms and audio books to the experimental and control groups and evaluated the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of preoperative audiobook application on blood pressure, pulse and anxiety levels of patients (Experimental): Patients in the experimental group will listen to an audio book for 20 minutes.
  Interventions: Other: audiobook app

INTERVENTIONS:
Other: audiobook app — audio book listening

SUMMARY:
Before the TDP surgery, the anxiety levels of the patients in the experimental group will be measured by listening to an audio book.

DETAILED DESCRIPTION:
Before Total Knee Prosthesis surgery, patients will have their blood pressure, pulse and anxiety levels measured before the surgery. Patients in the experimental group will listen to an audiobook for 20 minutes. The selected book will be played via wireless headphones. The researcher will check the battery level of the headphones and charge it when necessary. In this way, the headphones will be ready for the next patient. A smartphone with Spotify mobile application installed, which the researcher is a member of, will be used for the audiobook application. The connection between the headphones and the audiobook will be provided via Bluetooth. The patient will be present from the moment they start listening to the audiobook section, and if they experience any hearing problems or if there is an attempt to stop listening, immediate intervention will be made. Necessary interventions will be made for patients who experience interruptions during listening to listen again. After each application, the headphones will be cleaned with an antiseptic solution containing chlorhexidine 2%. The patient will be asked to rest for 10 minutes after the audiobook application. At the end of 10 minutes, the patient will be filled with an AÖKÖ and the patient's blood pressure and pulse will be measured and recorded. When measuring patients' blood pressure, the same blood pressure monitor with calibrated cuff, manometer, and stethoscope will be used, and when measuring pulse, the saturation device data will be used and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 40-80 years of age,
* Patients must be conscious and able to communicate,
* Individuals who volunteer to participate in the study,
* No hearing problems,
* Individuals who will undergo TKA surgery,
* Can understand Turkish,
* Patients must have elective (planned) surgery (must have been hospitalized at least 2 hours before surgery).

Exclusion Criteria:

* Refusing to participate in the study,
* Any communication barrier,
* Cancellation of TKA surgery for any reason.

Ages: 40 Months to 80 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The patients in the experimental and control groups consisted of male and female patients.
Enrollment: 70 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The Surgery Specific Anxiety Scale will be used for preoperative anxiety. | up to 12 months
  It was developed to determine the level of anxiety in surgical patients during and after surgery. The scale is a 5-point Likert-type scale consisting of 10 questions designed to measure the anxiety that patients may experience regarding surgery. The surgery-specific anxiety score in the scale is obtained by adding the responses to all items, and the total score of the scale is 50. As the score increases, the level of anxiety experienced also increases.
Patient Introduction Form | up to 12 months
  It consists of two parts. The first part includes introductory information such as the patient's age, gender, education level, and employment status, while the second part evaluates the total knee prosthesis surgery history, current chronic disease status, and knowledge about the audiobook. There will be a total of 10 questions in the form.
Patient Pulse Form, | up to 12 months
  Pulse findings of patients who will undergo total knee replacement surgery will be recorded before and after the audiobook application.
patient blood pressure form | up to 12 months
  Blood pressure findings of patients who will undergo total knee prosthesissurgery will be recorded before and after the audiobook application and it will be checked whether it is effective in reducing the blood pressure.

IPD SHARING:
Plan to Share IPD: No
ı don't know

REFERENCES:
- [Background] Sahin G, Basak T. The Effects of Intraoperative Progressive Muscle Relaxation and Virtual Reality Application on Anxiety, Vital Signs, and Satisfaction: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Jun;35(3):269-276. doi: 10.1016/j.jopan.2019.11.002. Epub 2020 Mar 4. PMID 32146074